CLINICAL TRIAL: NCT05030922
Title: Cardiovascular Risk Reduction-Diet in Pregnancy - Follow up 20 Years After the "CARRDIP"-Trial
Acronym: CARRDIP20
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Per Ole Iversen, MD (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Per Ole Iversen, MD, Professor, University of Oslo
Organization: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20/00301
Record Dates: First submitted 2021-08-20; First posted 2021-09-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet intervention (Experimental): Follow up of both mother and offspring 20 years after allocation to an antiatherogenic diet during pregnancy.
  Interventions: Other: Antiatherogenic diet
- Control (No Intervention): Follow up of both mother and offspring 20 years after allocation to control group during pregnancy.

INTERVENTIONS:
Other: Antiatherogenic diet — Participants instructed in antiatherogenic diet during pregnancy with frequent follow-ups to ensure compliance
  Arms: Diet intervention

SUMMARY:
The "Cardiovascular Risk Reduction-Diet in Pregnancy" (CARRDIP) - is a randomised controlled trial with dietary intervention during pregnancy. The participants were enrolled in Norway 20 years ago and consisted of 269 pregnant, healthy mothers. The participants were randomised 1:1 to either intervention-diet or control. The intervention diet was build upon an anti-atherogenic principle and was a so called "Mediterranean diet". The participants were monitored during pregnancy, and mother and child participated in a follow-up study 1 year after birth. The current "CARRDIP20" trial is a follow-up of the same participants, both mother and offspring, 20 years after the original intervention to measure and analyse the cardiovascular health and compare the intervention group to the control group.

ELIGIBILITY:
Inclusion Criteria from original CARRDIP-trial:

* Non-smoking pregnant women
* BMI 19 to 32 kg/m2 at inclusion
* Age 21 to 38 years
* Carrying a single foetus

Exclusion Criteria:

* Previous pregnancy complications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 538 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular health score | 1 day
  Cardiovascular risk score by use of the most appropriate available risk score algorithm available at time of analysis, at present the preferred calculator is Life's Simple 7 - The American Heart Association https://doi.org/10.1161/CIRCULATIONAHA.109.192703

SECONDARY OUTCOMES:
Blood samples - Lipid profile | 1 day
  Ratio of non-HDL cholesterol to HDL cholesterol in blood
Blood samples - Lipid profile | 1 day
  Lipoprotein a concentration in blood
Anthropometry | 1 day
  Waist-to-hip ratio (WHR)
Body fat percentage | 1 day
  Measured by bioimpedance
Ultrasound examination of liver | 1 day
  Ultrasound-Guided Attenuation Parameter (UGAP) of liver
Ultrasound examination of carotid artery | 1 day
  Intima-media thickness in carotid artery
Blood samples - Glukose metabolism | 1 day
  Hemoglobin A1c concentration in blood as a measure of long term blood sugar levels
Mean arterial pressure (MAP) | 1 day
  Measured by

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual patient data due to limitations in ethical approval and data protection considerations of the project.

REFERENCES:
- [Background] Khoury J, Haugen G, Tonstad S, Froslie KF, Henriksen T. Effect of a cholesterol-lowering diet during pregnancy on maternal and fetal Doppler velocimetry: the CARRDIP study. Am J Obstet Gynecol. 2007 Jun;196(6):549.e1-7. doi: 10.1016/j.ajog.2007.01.017. PMID 17547890
- [Background] Khoury J, Henriksen T, Christophersen B, Tonstad S. Effect of a cholesterol-lowering diet on maternal, cord, and neonatal lipids, and pregnancy outcome: a randomized clinical trial. Am J Obstet Gynecol. 2005 Oct;193(4):1292-301. doi: 10.1016/j.ajog.2005.05.016. PMID 16202717
- [Background] Khoury J, Henriksen T, Seljeflot I, Morkrid L, Froslie KF, Tonstad S. Effects of an antiatherogenic diet during pregnancy on markers of maternal and fetal endothelial activation and inflammation: the CARRDIP study. BJOG. 2007 Mar;114(3):279-88. doi: 10.1111/j.1471-0528.2006.01187.x. PMID 17217362
- [Derived] Troensegaard H, Khoury J, Westerberg AC, Tonstad S, Roeters van Lennep J, Veierod MB, Iversen PO, Holven KB, Retterstol K. Protocol for a 20-year follow-up after a randomized controlled trial of a Mediterranean diet in pregnancy: maternal and offspring risk factors for cardiovascular disease. Front Pediatr. 2023 Oct 18;11:1256815. doi: 10.3389/fped.2023.1256815. eCollection 2023. PMID 37920793
- See also: Link to project homepage on University of Oslo domain (norwegian) — https://www.med.uio.no/imb/forskning/prosjekter/hjertevennlig-kost-graviditet-langtidsoppfolging/